CLINICAL TRIAL: NCT04844723
Title: Pediatric Videolaryngoscopic Intubation and Difficult Airway Classification
Acronym: PeDiAC
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-10380-BO-ff
Record Dates: First submitted 2021-04-13; First posted 2021-04-14 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Airway Complication of Anesthesia; Intubation;Difficult; Anesthesia; Laryngoscopy; Airway Management
Keywords: Children; Airway management; Videolaryngoscopy; Endotracheal Intubation; Difficult Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study's primary aim is to develop and validate a multivariable diagnostic model for the prediction of difficult videolaryngoscopy (the 'PeDiAC classification') in children undergoing general anesthesia with tracheal intubation. The secondary aim is to compare the diagnostic performance of the PeDiAC-classification with the Cormack-Lehane classification.

DETAILED DESCRIPTION:
Difficult tracheal intubation is one of the major reasons for anesthesia-related adverse events. Videolaryngoscopy has become an important part of the anesthesiology standard of care for difficult airway management in the past decades. This is especially relevant in children, as their airway anatomy differs greatly from adults because they are likely incapable of tolerating brief apneic episodes. Still, medical preconditions and procedural and technical factors related to difficult videolaryngoscopy have not been broadly investigated and not fully been understood.

The primary aim of the PeDiAC study is to develop and validate a multivariable diagnostic model for the classification of difficult videolaryngoscopy (the 'PeDiAC classification') in children undergoing general anesthesia with tracheal intubation. Study planning and conduction are in accordance with the TRIPOD 'Transparent reporting of a multivariable prediction model for individual prognosis or diagnosis' statement. The secondary aim is to compare the diagnostic performance of the PeDiAC-classification with the Cormack-Lehane classification, which is the current clinical standard for assessing intubation via direct laryngoscopy. We conduct a prospective observational study that will include approximately 800 pediatric patients within one year scheduling for tracheal intubation. Patients with age below 18 years will be considered to be eligible for inclusion. Procedural and surgical data, as well as medical preconditions, will be assessed systematically. After tracheal intubation, performed by the responsible anesthetist, the intubation process will be rated by the responsible anesthetist and an additional independent observer, and detailed information regarding procedural and technical factors related to videolaryngoscopy will be documented. All sampled independent variables will be considered to be potential candidate predictors for the multivariable regression model.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing general anesthesia with tracheal intubation in the study center.
* Informed consent obtained
* Age < 18 years

Exclusion Criteria:

* Anesthetist prefers conventional laryngoscopy
* Indication for intubation via a bronchoscope or awake intubation

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Consecutive sampling: Pediatric patients undergoing general anesthesia with tracheal intubation in the study center.
Sampling Method: Non-Probability Sample
Enrollment: 809 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Difficult videolaryngoscopic intubation | 1 hour
  Rating by the responsible anesthetist

SECONDARY OUTCOMES:
First pass success rate | 1 hour
  Percentage of successful intubations with one attempt
Overall success rate with the first-choice technique | 1 hour
  Percentage of successful intubations without transition to another technique
Number of attempts | 1 hour
  Total number of laryngoscopy and intubation attempts until airway established
Change of airway technique | 1 hour
  Transition to a different technique, i.e. flexible bronchoscopy, surgical airway, supraglottic airway as clinically assessed (Yes/No)
Best glottic view | 1 hour
  Best view on the larynx obtained during laryngoscopy assessed by Cormack/Lehane classification (grade I to IV)
Time to best view | 1 hour
  Time until optimal view conditions during laryngoscopy
Intubation time | 1 hour
  Time until successful tracheal intubation
Intubation difficulty, ease of intubation and quality of visualisation | 1 hour
  Subjective ratings on visual analogue scales (0 to 100 with 0 being the best)
Post-intubation recommendation for an intubation method | 1 hour
  Requirement of recommendation for further intubations of the responsible anesthetist
Post-intubation recommendation for an anesthesia alert cart | 1 hour
  Recommendation of the responsible anesthetist (yes/no)
Post-intubation diagnosis of 'difficult intubation' | 1 hour
  Rating of the responsible anesthetist
Airway-related adverse events | 1 hour
  Laryngospasm, bronchospasm, larynx trauma, airway trauma, soft tissue trauma, oral bleeding, edema, dental damage, corticosteroid application, accidental esophageal intubation, aspiration, hypotension or hypoxia
Difficult bag-mask ventilation | 1 hour
  As clinically assessed (yes/no) by the responsible anesthetist
Lowest oxygen saturation | 1 hour
  Measured with pulsoxymetry during anesthesia
Hypercapnia | 1 hour
  Measured endtidal carbon dioxide after successful intubation

CONTACTS AND LOCATIONS:
Overall Officials: Martin Petzoldt, MD, Study Director — Universitätsklinikum Hamburg-Eppendorf; Thorsten W Dohrmann, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf; Christian Zöllner, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No